CLINICAL TRIAL: NCT04763876
Title: Comparison of Intramuscular Ketorolac at Two Single-Dose Regimens for Treatment of Acute Musculoskeletal Pain in a Military Emergency Department: A Randomized Controlled Non-Inferiority Trial
Brief Title: Intramuscular Ketorolac at Two Single-Dose Regimens
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: William Beaumont Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Edna Rath, Human Protections Director, William Beaumont Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C.2019.088
Record Dates: First submitted 2021-02-01; First posted 2021-02-21 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Musculoskeletal Pain; Analgesia; Adverse Event
Keywords: emergency department; ketorolac; musculoskeletal pain; non-inferiority; adverse event
MeSH Terms: conditions — Musculoskeletal Pain; Agnosia; Emergencies | interventions — Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Intervention Model Description: Single blinded, randomized, non-inferiority
Who Masked: Participant
Masking Description: The patient was unaware of the dosage of ketorolac they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 15 mg ketorolac intramuscular (Active Comparator): Patients who received a single 15 mg dose of ketorolac administered intramuscularly
  Interventions: Drug: Ketorolac Injection 15 mg
- 60 mg ketorolac intramuscular (Active Comparator): Patients who received a single 60 mg dose of ketorolac administered intramuscularly
  Interventions: Drug: Ketorolac Injection 60 mg

INTERVENTIONS:
Drug: Ketorolac Injection 15 mg — A single dose of 15 mg ketorolac administered intramuscularly.
  Other Names: toradol; ketorolac tromethamine; ketorolac
  Arms: 15 mg ketorolac intramuscular
Drug: Ketorolac Injection 60 mg — A single dose of 60 mg ketorolac administered intramuscularly.
  Other Names: Toradol; ketorolac tromethamine; ketorolac
  Arms: 60 mg ketorolac intramuscular

SUMMARY:
The purpose of this study was to evaluate a single 15 mg intramuscular (IM) dose of ketorolac for analgesic non-inferiority versus a single 60 mg IM dose for the treatment of acute MSK pain in a military emergency department (ED) that services Department of Defense (DoD), Department of Veteran Affairs (VA), and foreign military beneficiaries

DETAILED DESCRIPTION:
The primary purpose of this study is to evaluate a single 15 mg IM dose of ketorolac for analgesic non-inferiority versus a single 60 mg IM dose for the treatment of acute MSK pain in a military ED that services Department of Defense (DoD), Department of Veteran Affairs (VA), and foreign military beneficiaries. The authors chose to evaluate 15 mg rather than the previously identified 10 mg dose for ease of administration as ketorolac is manufactured in 15 mg/mL, 30 mg/mL, and 60 mg/2mL vials in the U.S. The dose of ketorolac served as the primary independent variable for the study and the change in Visual Analog Scale (VAS) score served as the dependent variable. Prescribing the minimally effective doses of NSAIDs is pertinent to prevent and reduce the number of adverse events. Thus, the secondary outcome assessed for the dose-dependence of subjective and objective adverse events with ketorolac.

ELIGIBILITY:
Inclusion Criteria:

* Tricare beneficiaries between 18-55 years of age
* Triaged as Emergency Severity Index 4 or 5
* Presenting to the William Beaumont Army Medical Center Emergency Department with a chief complaint of acute MSK pain (i.e., general muscular, neck, back, shoulder, arm, forearm, elbow, wrist, finger, hip, knee, thigh, leg, ankle, foot, or digits)
* Pain intensity of 20 mm or greater on a standard 100 mm visual analog scale
* Who the attending provider concurred with ketorolac IM administration for analgesia.

Exclusion Criteria:

* Body weight less than 50 kg (110 lbs.)
* Younger than 18 or older than 55 years
* Pregnant or breast feeding
* History of: confirmed, unconfirmed, known, unknown, or suspected peptic ulcer disease, intestinal hemorrhage, renal insufficiency, hepatic insufficiency, cerebrovascular bleeding, hemorrhagic diathesis, incomplete hemostasis, dark stools, bright red blood per rectum, hemoptysis, easy bruising, or high risk of bleeding
* Unable to confidently convey or unknown medical history
* Allergy or hypersensitivity to nonsteroidal anti-inflammatory drugs or aspirin
* Systolic blood pressure <90 or >180 mmHg
* Pulse rate <50 or >150 beats/min
* Any over-the-counter or prescribed opioid and/or non-opioid analgesic medication (oral, per rectum, topical or parenteral) taken within 12 hours of ED presentation
* Advised by any medical provider to not receive NSAIDs for any reason
* Pain duration greater than 30 days (including acute on chronic pain)
* Refusal to remain in the WBAMC ED for up to 60 minutes after injection of ketorolac
* Patients currently taking anticoagulant medications
* Concurrent use of medications which are contraindicated with concomitant NSAID use (drugs include aspirin, probenecid and pentoxifylline).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2020-06-27 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2021-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel J Turner, MPAS, Principal Investigator — Department of Emergency Medicine, William Beaumont Army Medical Center
Locations (1):
- William Beaumont Army Medical Center, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For the duration of our study, no study subjects were excluded or disenrolled.
Period: Overall Study
Arm/Group | 15 mg Ketorolac Intramuscular | 60 mg Ketorolac Intramuscular
Started | 55 | 55
Completed | 55 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 15 mg Ketorolac Intramuscular | 60 mg Ketorolac Intramuscular | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 14 | 31
  Between 18 and 65 years | 38 | 41 | 79
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 31.1 [19 to 51] | 30.7 [18 to 54] | 30.9 [18 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 30
  Male | 42 | 38 | 80
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 55 | 55 | 110
Weight in kilograms [Mean (Full Range); unit: kg] | 82.8 [51 to 135] | 84.5 [53 to 131] | 83.7 [51 to 135]
Duration of pain [Mean (Full Range); unit: minutes] | 69.8 [31 to 100] | 66.3 [24.8 to 100] | 68 [24.8 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference of Visual Analog Scale Scores
Description: The mean difference of Visual Analog Scale scores between the two treatment groups measured at 60-minutes. The Visual Analog Scale used measures from 0 mm to 100mm. A higher score represents more degree of change. 13 mm was used as the non-inferiority margin. A difference between the two groups less than 13 mm demonstrates that 15 mg is non-inferior to 60 mg.
Time Frame: 60 minutes from administration of medication
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 15 mg Ketorolac Intramuscular | 60 mg Ketorolac Intramuscular
Number analyzed (Participants) | 55 | 55
score on a scale | -29.74 (22.46) | -29.85 (23.14)

2. Secondary Outcome: Mean Difference of Visual Analog Scale Scores
Description: The mean difference of Visual Analog Scale scores between the two treatment groups measured at 30-minutes. The Visual Analog Scale used measures from 0 mm to 100mm. A higher score represents more degree of change. 13 mm was used as the non-inferiority margin. A difference between the two groups less than 13 mm demonstrates that 15 mg is non-inferior to 60 mg.
Time Frame: 30 minutes from administration of medication
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 15 mg Ketorolac Intramuscular | 60 mg Ketorolac Intramuscular
Number analyzed (Participants) | 55 | 55
score on a scale | -18.99 (17.73) | -17.31 (18.31)

3. Secondary Outcome: Number of Participants With Adverse Events Related to the Administration of Ketorolac
Description: The incidence of observed objective and reported subjective adverse events related to the administration of ketorolac.
Time Frame: At time of administration, 30 minutes after administration, and 60 minutes after administration.
Measure: Count of Participants; unit: Participants
Arm/Group | 15 mg Ketorolac Intramuscular | 60 mg Ketorolac Intramuscular
Number analyzed (Participants) | 55 | 55
Participants | 1 | 9

ADVERSE EVENTS:
Time Frame: 120 minutes
Arm/Group | 15 mg Ketorolac Intramuscular | 60 mg Ketorolac Intramuscular
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 1/55 | 9/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15 mg Ketorolac Intramuscular (N=55) | 60 mg Ketorolac Intramuscular (N=55)
Burning at site of injection (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Fatigue (Nervous system disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT04763876/Prot_001.pdf
  • Statistical Analysis Plan (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT04763876/SAP_000.pdf
  • Informed Consent Form (2020-03-13): https://cdn.clinicaltrials.gov/large-docs/76/NCT04763876/ICF_002.pdf